CLINICAL TRIAL: NCT06487208
Title: AnticipaMax: Impact of the Use of a Hand-held Digital Cognitive Aid in Order to Anticipated a Potential Crisis Situation, Measured by a Composite Globale Performance Score, in Anesthesia Resident
Brief Title: Impact of a Hand-held Digital Cognitive Aid to Anticipated a Simulated Crisis Situation for Resident
Acronym: AnticipaMax
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Principal Investigator, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AnticipaMax
Record Dates: First submitted 2024-06-14; First posted 2024-07-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Anticipation; Cognitive aid; Critical situation; Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): No intervention
  Interventions: Other: Placebo
- AnticipaMax (Experimental): The subjects will be instructed to use the 5 minutes to consider potential complications, prioritize them, and anticipate their management. The facilitators will have a neutral role with pre-determined standardized responses and will ensure the correct use of the Max tool during this time period
  Interventions: Other: Use of a digital cognitive aid in order to anticipate a critical situation

INTERVENTIONS:
Other: Use of a digital cognitive aid in order to anticipate a critical situation — Use of a digital cognitive aid in order to anticipate a critical situation
  Arms: AnticipaMax
Other: Placebo — No intervention
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate that the systematic anticipation of major potential per operative complications using a digital cognitive aid and visualizing the appropriate actions in such cases leads to an improvement in overall performance during an immediate critical situation in simulation, particularly through the regular reassessment of the initial hypothesis

DETAILED DESCRIPTION:
Context: Over the past few decades, considerable efforts have been made to understand and manage risks, especially in high stakes sectors such as aviation and the nuclear industry. However, risk management in the medical field, such as anesthesia and critical care, is still in its infancy. Complex activities like anesthesia and critical care are prone to human errors, exacerbate by factors such as lack of sleep and stress.

Despite the inevitable risk of errors, solution exist to reduce them, including the use of cognitive aids such as the digital application MAX or the SFAR paper checklists. The value of these aids is well documented and supported by extensive literature. Nevertheless, those tools are still underutilized in clinical practice, likely due to negative perceptions and, a lack of familiarity among doctors.

Thus, the investigators believe that the systematic anticipation of perioperative complications and their management through a digital cognitive aid in daily practice could improve patient care by enhancing the overall performance of doctors and healthcare teams.

Primary objective: Demonstrate that the systematic anticipation of potential major perioperative complications, by using a digital cognitive aid, improves global performance in managing a critical situation. The primary outcome is measure with a composite score including both technical and no technical performance.

Secondary objectives: Several secondary outcomes measures: Comparison between the two groups of the technical and no technical performance. Stress during the simulation, self confidence level, the difference between the required competency level and the level that participant estimates have. And evaluation of biological stress response through sympathetic and parasympathetic indices calculated from electrophysiological variables via a connected watch.

Nature and conduct of the study: A prospective, randomized, controlled, single center study (Lyon). The study will be conducted in simulation at CLESS (Claude Bernard University Lyon 1) with participants being anesthesia and critical care residents in the consolidation and advanced phases. A single scenario will be used for the study. Each resident will be randomized into either the interventional group (anticipaMAX) or the control group. The intervention will take place during the five minutes preceding the start of the scenario. During this period, volunteers in the interventional group will be instructed to use the five minutes to consider potential complications and anticipate their management with the help of the MAX tool. Volunteers in the control group will be free to organize themselves as they wish, with the same medical file elements and the MAX application at their disposal. During the scenario, facilitator intervention will be standardized to ensure the comparability between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia Resident of Lyon

Exclusion Criteria:

* First Year of anesthesia residency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Global performance composite score | one day after simulation
  The primary outcome measure is a composite score of overall performance, based on both technical performance and non-technical performance, assessed by a validated scale (Ottawa Crisis Resource Management) demonstrated by the included subject during the full-scale simulation after the implementation of the intervention.
  Composite score of technical performance on a scale of 100 + non-technical performance on a scale of 0 minimum to a maximum of 100, therefore a total from zero minimum to 200 hundred maximum.
  To obtain this composite score, we will sum the technical performance score out of 100 points and the non-technical performance score out of 100 points (Ottawa scale / 42 points, converted to a score out of 100).

SECONDARY OUTCOMES:
Technical performance | One day after simulation
  performance score from 0 minimum to a maximum of 100
Non technical performance | One day after simulation
  performance score from 0 minimum to a maximum of 100
Stress level, self-evaluated | 2 minutes before simulation
  Visual analog scale from 0 minimum to 100 maximum
Stress level, self-evaluated | 2 minutes after simulation
  Visual analog scale from 0 minimum to 100 maximum
Self confidence level | 2 minutes after simulation
  Visual analog scale from 0 minimum to 100 maximum
Difference between the required competency level and the level that participant estimates have | 2 minutes after simulation
  Visual analog scale from 0 minimum to 100 maximum

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Cejka, Ph.D, Study Director — Université Claude Bernard Lyon 1
Locations (1):
- HENKEME Mathieu, Lyon, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Background] Evain JN, Perrot A, Vincent A, Cejka JC, Bauer C, Duclos A, Rimmele T, Lehot JJ, Lilot M. Team planning discussion and clinical performance: a prospective, randomised, controlled simulation trial. Anaesthesia. 2019 Apr;74(4):488-496. doi: 10.1111/anae.14602. Epub 2019 Feb 15. PMID 30768684
- [Background] Paraschiv AP, Balanca B, Lilot M, Aigle L, Lehot JJ, Cejka JC. Use of a Digital Cognitive Aid Improves Memorization of Military Caregivers After High-Fidelity Simulations of Combat Casualty Care. Mil Med. 2023 Jan 4;188(1-2):e295-e300. doi: 10.1093/milmed/usab175. PMID 33928372
- [Background] Truchot M, Balanca B, Wey PF, Tazarourte K, Lecomte F, Le Goff A, Leigh-Smith S, Lehot JJ, Rimmele T, Cejka JC. Use of a Digital Cognitive Aid in the Early Management of Simulated War Wounds in a Combat Environment, a Randomized Trial. Mil Med. 2020 Aug 14;185(7-8):e1077-e1082. doi: 10.1093/milmed/usz482. PMID 32091610
- [Background] Claverie D, Trousselard M, Sigwalt F, Petit G, Evain JN, Bui M, Guinet-Lebreton A, Chassard D, Duclos A, Lehot JJ, Rimmele T, Canini F, Lilot M. Impact of stress management strategies and experience on electrodermal activity during high-fidelity simulation of critical situations. Br J Anaesth. 2020 Nov;125(5):e410-e412. doi: 10.1016/j.bja.2020.07.024. Epub 2020 Aug 21. No abstract available. PMID 32838978
- [Background] Lelaidier R, Balanca B, Boet S, Faure A, Lilot M, Lecomte F, Lehot JJ, Rimmele T, Cejka JC. Use of a hand-held digital cognitive aid in simulated crises: the MAX randomized controlled trial. Br J Anaesth. 2017 Nov 1;119(5):1015-1021. doi: 10.1093/bja/aex256. PMID 29028930